CLINICAL TRIAL: NCT03647163
Title: Phase 1-2 Trial of Systemically Administered VSV-IFNβ-NIS in Combination With Checkpoint Inhibitor Therapy in Patients With Selected Solid Tumors
Brief Title: Ph I/II Trial of Systemic VSV-IFNβ-NIS in Combination With Checkpoint Inhibitor Therapy in Patients With Select Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vyriad, Inc. (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VYR-VSV2-202
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor; Non Small Cell Lung Cancer; Neuroendocrine Carcinoma; Renal Cell Carcinoma (RCC)
Keywords: NSCLC; NEC; RCC; Non-small cell lung cancer; Neuroendocrine; Renal Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Neuroendocrine; Carcinoma, Renal Cell | interventions — pembrolizumab; Ipilimumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: Safety run-in with dose escalation to be used to identify the optimum dose for expansion. Dose expansion will recruit patients in parallel into 3 groups, NSCLC, NEC and RCC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Safety Run-in Dose Level 1 (Experimental): Patients with pembrolizumab refractory solid tumors will receive a single IV dose of 5e10 TCID50 VSV-IFNβ-NIS in combination with Pembrolizumab at standard labeled dose administered on day 1, then every 21 days, up to 2 years.
  Interventions: Biological: VSV-IFNβ-NIS; Biological: Pembrolizumab
- Safety Run-in Dose Level 2 (Experimental): Patients with pembrolizumab refractory Neuroendocrine Carcinoma (NEC) or non small cell lung cancer (NSCLC) will receive a single IV dose of 1.0e11 TCID50 VSV-IFNβ-NIS in combination with Pembrolizumab at standard labeled dose administered on day 8, then every 21 days, up to 2 years.
  Interventions: Biological: VSV-IFNβ-NIS; Biological: Pembrolizumab
- Expansion NEC (Experimental): Patients with pembrolizumab refractory Neuroendocrine Carcinoma (NEC) will receive a single IV dose of 1.0e11 TCID50 VSV-IFNβ-NIS in combination with Pembrolizumab at standard labeled dose administered on day 8, then every 21 days, up to 2 years.
  Interventions: Biological: VSV-IFNβ-NIS; Biological: Pembrolizumab
- Expansion NSCLC arm (Experimental): Patients with pembrolizumab refractory non small cell lung cancer (NSCLC) will receive a single IV dose of 1.0e11 TCID50 VSV-IFNβ-NIS in combination with Pembrolizumab at standard labeled dose administered on day 8, then every 21 days, up to 2 years.
  Interventions: Biological: VSV-IFNβ-NIS; Biological: Pembrolizumab
- Expansion Part D (Experimental): Patients with non small cell lung cancer (NSCLC) or Neuroendocrine Carcinoma (NEC) will receive a single IV dose of VSV-IFNβ-NIS on Day 4 in combination with ipilumumab + nivolumab at standard labeled dose administered on Day 1 then every 21 days up to 2 years.
  Interventions: Biological: VSV-IFNβ-NIS; Biological: ipilimumab + nivolumab
- Expansion Renal Cell Carcinoma (RCC) Part E (Experimental): Arm Description: Renal Cell Carcinoma (RCC) will receive a single IV dose of VSV-IFNβ-NIS on Day 4 in combination with ipilumumab + nivolumab at standard labeled dose administered on Day 1 then every 21 days for a total of 4 Cycles. Nivo Single agent will be administered every 28 days starting with Cycle 5 for a total treatment period of up to 2 years.
  Interventions: Biological: VSV-IFNβ-NIS; Biological: ipilimumab + nivolumab

INTERVENTIONS:
Biological: VSV-IFNβ-NIS — Intravenous oncolytic Vesicular stomatitis virus (VSV) expressing Interferon-beta (IFNβ) and the sodium iodide symporter (NIS)
  Other Names: Voyager-V1; VSV; VSV2
Biological: Pembrolizumab — Pembrolizumab
  Arms: Expansion NEC; Expansion NSCLC arm; Safety Run-in Dose Level 1; Safety Run-in Dose Level 2
Biological: ipilimumab + nivolumab — Intravenous ipilimumab 1mg/kg in combination with nivolumab 360mg, or Intravenous ipilimumab 1mg/kg in combination with nivolumab 3mg/ kg for 4 cycles, followed by fixed dose nivolumab 480mg
  Arms: Expansion Part D; Expansion Renal Cell Carcinoma (RCC) Part E

SUMMARY:
The safety run-in portion of this study is designed to identify the optimal dose of VSV-IFNβ-NIS in combination with pembrolizumab in patients with solid tumors and follows the 3+3 design. The expansion portion will use one-sample binomial designs to assess the efficacy of the combination in patients with refractory NSCLC or NEC. The optimal dose (RP2D) determined in the dose escalation portion of the trial will be used for the expansion portion. The study has been conducted with a dose of 1.7 × 1010 as the recommended phase II dose in an expansion cohort of 10 patients with NSCLC. However, current data suggests that VSV-IFNβ-NIS doses of up to 1.7 × 1011 is safe and likely more efficacious. Thus, this study will test a second VSV-IFNβ-NIS dose level, 1.0x1011 TCID50. A safety assessment will be carried out after 3 patients are enrolled. If this dose schedule is well tolerated and virus PK are not negatively impacted, both the NSCLC and NEC expansion cohorts will open using this dose schedule. If 2 of the first 3 patients or 2 of the first 6 patients experience a DLT, the dose will be de-escalated to 5 x 1010. The safety run-in/dose escalation portion of this study is expected to require a minimum of 3 patients and a maximum of 18 patients (6 patients per dose level). The expansion portion of this study is expected to require a minimum of 10 per cohort. The NSCLC and NEC patients enrolled at the identified optimal dose in the dose escalation cohort would be included in the dose expansion cohort if they are evaluable for the primary endpoint in the expansion portion (4 dose escalation patients at the optimal dose are expected to roll over to the expansion). Additionally, up to 16 Renal Cell Carcinoma (RCC) patients will be treated in the expansion cohort. This will permit up to 86 treated patients.

DETAILED DESCRIPTION:
All patients will be dosed with VSV-IFNβ-NIS on day 1. For Part A, Part B [Group 1], and Part C [Group 1] pembrolizumab will be administered on day 1 (concurrent pembrolizumab dosing). For Part A, and Parts B and C [Group 2] pembrolizumab may be administered on day 8 (delayed pembrolizumab dosing). pembrolizumab treatment will continue Q3W per the Keytruda® USPI, with efficacy evaluations after cycle 2 then every 9 weeks until PD.

In Part D, NSCLC and NEC patients will be dosed with Nivo + ipi on Cycle 1 Day 1 and with VSV-IFNβ-NIS on day 4 (single dose). Nivo + ipi will continue to be given Q3W with efficacy evaluations at Cycle 3 and every 9 weeks thereafter.

In Part E, RCC patients will be dosed with Nivo + ipi on Cycle 1 Day 1 and with VSV-IFNβ-NIS on day 4 (single dose). Nivo + ipi will continue to be given Q3W for 4 cycles, then Nivolumab monotherapy Q4W fixed dose of 480mg. Efficacy assessments will be performed Q9W.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of:

  * Arm 1: dose level 1 and below: Advanced and/or metastatic solid tumors for which no existing options are felt to provide clinical benefit
  * Arm 2: dose level 2: Advanced and/or metastatic NSCLC OR NEC in which radiological progression has been demonstrated during therapy with a PD-1/PD-L1 immune checkpoint inhibitor, and for which no existing options are felt to provide clinical benefit.
  * Arm 3: Advanced and/or metastatic NEC in which radiological progression has been demonstrated during therapy with a PD-1/PD-L1 immune checkpoint inhibitor, and for which no existing options are felt to provide clinical benefit.
  * Arm 4: Advanced and/or metastatic NSCLC in which radiological progression has been demonstrated during therapy with a PD-1/PD-L1 immune checkpoint inhibitor, and for which no existing options are felt to provide clinical benefit.
  * Arm 5: NEC: poorly differentiated NEC (large or small cell, or not further specified) with progressive disease following at least one prior line of systemic therapy.
  * Arm 6: RCC: histologically confirmed diagnosis of advanced or metastatic RCC, including all IMDC risk categories (favorable, intermediate, and poor risk).
* Measurable disease based on RECIST 1.1. The first 3 patients in the safety run-in phase do not need measurable disease. Part C: advanced NEC (neuroendocrine carcinoma based on histopathology according to WHO criteria. Patients with small cell carcinoma, large cell neuroendocrine carcinoma, and neuroendocrine carcinoma not otherwise specified, of any primary organ are eligible in which radiological progression has been demonstrated during therapy with a PD-(L)1 immune checkpoint inhibitor, and for which no existing options are felt to provide clinical benefit.
* Performance status of 0 or 1 on the ECOG Performance Scale.
* Life expectancy of >3 months if not on active anti-cancer therapy
* Willingness to provide biological samples required for the duration of the study including a fresh tumor biopsy sample.
* Adequate organ function using predefined laboratory values obtained ≤14 days prior to registration.
* Negative pregnancy test for female patients of childbearing potential
* Absence of active CNS involvement. NOTE: Pre-enrollment imaging of asymptomatic patients not mandatory
* Ability to provide written informed consent.
* Willing and able to comply with scheduled visits, treatment schedule, and laboratory testing.

Exclusion Criteria:

* Availability of and patient acceptance of curative therapy.

  a. For NSCLC cohort: i. Known EGFR mutations which are sensitive to available targeted inhibitor therapy (including, but not limited to, deletions in exon 19 and exon 21 [L858R] substitution mutations). All patients with non-squamous histology must have been tested for EGFR mutation status; use of an FDA-approved test is strongly encouraged. ii. Non-squamous histology and unknown or indeterminate EGFR status. b. Part D NSCLC cohort: Known ALK translocations which are sensitive to available targeted inhibitor therapy. If tested, use of an FDA-approved test is strongly encouraged. Patients with unknown or indeterminate ALK status may be enrolled.
* Recent or ongoing serious infection, including:

  1. Any active Grade 3 or higher (per the NCI CTCAE, version 4.03) viral, bacterial, or fungal infection within 2 weeks of registration.
  2. Known seropositivity for or active infection by the human immunodeficiency virus (HIV).
  3. Acute hepatitis B or acute hepatitis C. Patients with chronic hepatitis B or hepatitis C may be enrolled provided their liver function is adequate as per section 3.17
  4. Known history of active TB (Bacillus tuberculosis).
* Any serious health condition, which, in the opinion of the investigator, would place the patient at undue risk from the study, including uncontrolled hypertension and/or diabetes, clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease requiring hospitalization within 3 months) or neurological disorder (e.g., seizure disorder active within 3 months)
* Prior therapy within the following timeframe before the planned start of study treatment as follows:

  * Chemotherapy, small molecule inhibitors, radiation, interventional radiology procedure, and/or other investigational agent: ≤3 weeks or 5 half-lives, whichever is shorter
  * Other monoclonal antibodies, antibody-drug conjugates, radioimmunoconjugates, or experimental therapies: ≤4 weeks (≤3 weeks with documented disease progression)
  * Prior palliative radiotherapy to non-CNS lesions must have been completed at least 2 weeks prior to randomization. Subjects with symptomatic tumor lesions at baseline that may require palliative radiotherapy within 4 weeks of randomization are strongly encouraged to receive palliative radiotherapy prior to randomization.
  * NSCLC patients only: prior chemotherapy or immunotherapy or a combination of chemotherapy and immunotherapy for stage IV NSCLC.
  * RCC patients:

    i. Previously received a CTLA-4 inhibitor in the first-line setting. ii. Relapsed/progressed during adjuvant immunotherapy with a PD-(L)1 inhibitor or relapse within 12 months after completion of adjuvant immunotherapy
* New York Heart Association classification III or IV, known symptomatic coronary artery disease, or symptoms of coronary artery disease on systems review, or known cardiac arrhythmias (atrial fibrillation or SVT) (Appendix II).
* Any known or suspected active organ-threatening autoimmune disease, such as inflammatory bowel disease, autoimmune hepatitis, lupus, or pneumonitis, with the exception of hypothyroidism and type 1 diabetes that are controlled with treatment.
* Immunodeficiency or immunosuppression, including systemic corticosteroids at >10mg/day prednisone or equivalent within 1 week prior to planned start of study treatment
* History of severe immune-mediated adverse reaction to immune checkpoint inhibitors.
* Toxicities from previous therapies that have not resolved to a grade 1 or less.
* History of non-infectious pneumonitis that required steroids, or current pneumonitis, or carcinomatous meningitis, or interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
* High volume disease, as assessed clinically via parameters such as radiologic impression and tumor markers or LDH.
* Portal vein thrombosis involving more than intrahepatic portal vein branches: thrombosis of the right or left portal vein branch or the bifurcation, partial or complete obstruction of the portal vein trunk.
* Known concurrent malignancy that is progressing or requires active treatment. EXCEPTIONS: basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in-situ cervical cancer that has been treated with curative intent, prostate cancer confined to the prostate gland with Gleason score <6 or PSA <1, as well as any stage I cancer treated with curative intent or any prior cancer with a disease-free interval of ≥3 years.
* Other concurrent anti-cancer therapy (chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (used for a non-FDA approved indication and in the context of a research investigation)).
* Neuroendocrine neoplasms described as "well-differentiated" or "moderately differentiated" on pathologic review, or reported as "carcinoid", i.e., not true poorly differentiated neuroendocrine carcinoma [Nagtegaal 2020].
* Has received a live vaccine within 30 days of planned start of study treatment. Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines and are NOT allowed.
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women or women of reproductive ability who are unwilling to use highly effective contraception
  * Nursing women
  * Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 4 weeks after stopping treatment.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Expansion arms: Overall response rate (ORR) | 43 days - 6 months
  proportion of patients in the analysis population who have complete response (CR) or partial response (PR) based on RECIST 1.1 imaging
Safety run-in arm: Number of participants with treatment related adverse events (NCI CTCAE; Version 4.03) | 21 days
  Assessment of safety and toxicity of intravenous VSV-IFNβ-NIS in combination with pembrolizumab therapy

SECONDARY OUTCOMES:
Overall Survival (OS) | 6 months
  Survival time is defined as the time from registration to death due to any cause.
Progression Free Survival (PFS) | 6 months
  Progression-free survival is defined as the time from registration to the earliest date documentation of disease progression or death due to any cause
Duration of response | 6 months
  defined for all evaluable patients who have achieved an objective response as the date at which the patient's earliest best objective status is first noted to be either a CR or PR to the earliest date progression is documented.
Disease Control Rate (DCR) | 6 months
  proportion of patients in the analysis population who have complete response (CR), partial response (PR) or stable disease (SD) based on RECIST 1.1 imaging on day 43.
Adverse events | 6 months
  All eligible patients that have initiated treatment will be considered evaluable for assessing adverse event rate(s). The maximum grade for each type of adverse event will be recorded for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Adjei, MD, PhD, Principal Investigator — The Cleveland Clinic; Patrick McGarrah, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No